CLINICAL TRIAL: NCT04135118
Title: Prospective Validation of a Prediction Model for Diagnosing Adenomyosis With Ultrasound.
Brief Title: Validation of the Adenomyosis Calculator
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: The Hospital of Vestfold (Other); University Hospital, Akershus (Other); St. Olavs Hospital (Other); Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Marit Lieng, Head of department, dept. of gynecology, Oslo University Hospital, Oslo University Hospital
Other Study IDs: OUS P360
Record Dates: First submitted 2019-10-16; First posted 2019-10-22 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Adenomyosis; Pelvic Pain Syndrome
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Adenomyosis is a disease where ectopic endometrial glands affect the muscular wall of the uterus. Women that suffer from dysmenorrhea or infertility caused by adenomyosis need to confirm or rule out adenomyosis, and therefore tools for non-histologic confirmation of adenomyosis are indubitably required. Transvaginal ultrasound has been shown to be useful in diagnosing adenomyosis, but the interpretation of findings requires significant expertise in ultrasound and experience with diagnosing adenomyosis. This is because adenomyosis shows a very heterogeneous appearance in ultrasound. There are many different diagnostic signs that have to be considered and weighed.

In a previous study, the investigators have developed a diagnostic algorithm that helps clinicians diagnose adenomyosis with transvaginal ultrasound and a clinical examination. It showed good diagnostic accuracy and seemed to be very robust with regards to artifacts and experience of the examiner. It is now necessary to validate this prediction model in a new, prospective study so it can be used in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal (defined by having had menstruation the last six month)
* If amenorrhea with levonorgestrel intrauterine device, the woman should be < 45 years old
* Hysterectomy planned due to a benign condition
* Hysterectomy does not require morcellation it is allowed to divide the uterus into 2-3 pieces, given that the orientation of the specimen is still possible for the pathologist)
* Written consent is given
* Can communicate in Norwegian or English at the Norwegian study sites, and Finnish, Swedish or English at the Finnish study site.

Exclusion Criteria:

* Gynecological cancer present at the time of inclusion
* Use of gonadotropin-releasing hormone agonist or antagonist within the last 3 months prior to the ultrasound evaluation
* Prior endometrial ablation or resection
* Postmenopausal status or no menstrual bleeding for the last 6 months, or amenorrhea with levonorgestrel-intrauterine device and age >45 years.
* Need for morcellation of the uterus

Max Age: 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A consecutive sample of women that are scheduled for a hysterectomy at one of the study sites and fulfill eligibility criteria are invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the prediction model for adenomyosis | 1 year
  Diagnostic accuracy will be described using sensitivity (in %), specificity (in %), positive predictive value (in %), negative predictive value (in %), positive likelihood ratio (calculated by sensitivity/1-specificity), negative likelihood ratio (calculated as 1-sensitivity/specificity) and the area under the receiver-operator curve (as calculated with the (0-1) of the model.

SECONDARY OUTCOMES:
Intraclass correlation coefficient (ICC) between readers | 2 years
  ICC values are categorized as follows: 0-0.20, slight agreement; 0.21-0.40, fair agreement; 0.41-0.60, moderate agreement; 0.61-0.80, substantial agreement; and 0.81-1, almost perfect agreement

CONTACTS AND LOCATIONS:
Overall Officials: Marit Lieng, Phd, Principal Investigator — Oslo University Hospital, Oslo, Norway
Locations (5):
- Turku University Hospital, Turku, Finland
- Norway (4):
  - Akershus University Hospital, Dept. of gynecology, Lørenskog, Akershus
  - St. Olavs Hospital, Dept. of Gynecology, Trondheim, Trøndelag
  - Sykehuset i Vestfold, Tønsberg, Vestfold
  - Department of Gynecology, Oslo University Hospital Ullevål and Rikshospital, Oslo

IPD SHARING:
Plan to Share IPD: Yes
We will share the values of all evaluated predictors in the model so that they can be used for re-calculation.
Supporting Information: Study Protocol, SAP
Time Frame: The data is planned to be made available within a year after the publication of all results.
Access Criteria: Access will be granted upon request and evaluation of the intended use of the data. The intended use should primarily gain improved patient care and research into adenomyosis and a detailed protocol has to be submitted.

REFERENCES:
- [Background] Tellum T, Nygaard S, Skovholt EK, Qvigstad E, Lieng M. Development of a clinical prediction model for diagnosing adenomyosis. Fertil Steril. 2018 Oct;110(5):957-964.e3. doi: 10.1016/j.fertnstert.2018.06.009. PMID 30316443